CLINICAL TRIAL: NCT05081999
Title: De-Adoption βeta-Blockers in Patients With Stable Ischemic Heart Disease Without REduced LV Ejection Fraction, Ongoing Ischemia, or Arrhythmias: a pragmaTic randomizEd Trial With Blinded Endpoints
Brief Title: De-Adoption of Beta-Blockers in Patients With Stable Ischemic Heart Disease
Acronym: ABBREVIATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00113192
Record Dates: First submitted 2021-09-20; First posted 2021-10-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Stable Ischemic Heart Disease; Coronary Artery Disease; Beta-blocker Therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Independent Medical Evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuation of Beta-Blockers (Other): For patients already on β-blocker therapy, the treatment will be continued and titrated at the discretion of the patient's most responsible physician(s).
  Interventions: Other: Medical Assessment; Other: Quality of Life Assessment
- De-Adoption of Beta-Blockers (Other): For patients on β-blocker therapy, medication will be tapered over 3-7 days to minimize the potential for withdrawal-related symptoms. A standardized angina treatment algorithm, which is independent of β-blocker use, will minimize any worsening of angina symptoms during drug withdrawal by utilizing other guideline recommended anti-anginal agents, such as calcium-channel blockers, long acting nitrates, or ivabradine. An anticipated 5% of patients allocated to this arm will not be able to tolerate discontinuation, however, patients will continue participation as per intention-to-treat principle. Background lifestyle measures and medical therapies will be recommended according to current Canadian guideline recommendations and individual patient profiles. Structured algorithms to achieve blood pressure goals that exclude the use of a β-blocker based on the Canadian Hypertension Education Program Guidelines will be provided.
  Interventions: Other: Medical Assessment; Other: Quality of Life Assessment

INTERVENTIONS:
Other: Medical Assessment — medical hx, events inquiry, adherence to treatment arm periodically over 4 years
Other: Quality of Life Assessment — online questionnaires periodically over 4 years, including SAQ, EQ-5D-5L, IIEF-5 (males) or FSFI (females)

SUMMARY:
Patients with heart disease are often prescribed many medications and these patients may experience drug interactions or negative drug related side effects. With newer medications and treatments available, it is not well known whether older drugs, such as beta-blockers, are still an effective and safe option for treating heart disease. Some evidence suggests beta-blockers should be continued, whereas other evidence suggests beta-blockers might cause unnecessary harm. The study hopes to determine whether continuation or discontinuation of beta-blockers will affect long term cardiovascular outcomes. The study investigators will also examine how beta-blockers continuation or discontinuation affects several quality of life measures.

DETAILED DESCRIPTION:
Patients will be randomized to continue β-blocker therapy or discontinue β-blocker therapy. Patients will be followed remotely for approximately four years for adherence, events and outcomes assessments, and completion of multiple web-based quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 years
2. Documented Coronary Artery Disease (CAD) defined as:

   * Myocardial Infarction at least 6 months prior; or
   * Stable ischemic heart disease (defined using one of the following tests suggestive of significant coronary artery disease):

     i. Positive exercise stress test ii. Positive Nuclear perfusion scan iii. Positive exercise or pharmacologic echocardiographic stress test iv. Positive magnetic resonance imaging coronary perfusion scan v. Coronary computed tomographic angiography Angiogram with stenosis ≥ 70% (or left main coronary artery ≥ 50%) or significant function disease based or positive fractional flow reserve testing by CT (FFRCT); vi. Invasive coronary angiography with ≥ 70% (or left main coronary artery ≥ 50%) or significant function disease based or positive fractional flow reserve testing (FFR) or instant wave free ratio (IFR),
   * Previous Percutaneous Coronary Intervention (PCI, at least 6 months prior if revascularization is performed for an MI); or
   * Previous Coronary Artery Bypass Grafting (CABG, at least 6 months prior if revascularization is performed for an MI)
3. Able and willing to provide informed consent

Exclusion Criteria:

1. Left Ventricular Ejection Fraction < 40% or current hospitalization for heart failure
2. Myocardial infarction <6 months prior to randomization
3. Indication for β-blocker as determined by the treating physician (such as atrial or ventricular arrhythmias or ongoing angina not controlled by another agent)
4. Uncontrolled hypertension or uncontrolled angina symptoms (per the Investigator's discretion)
5. Non-compliance with medical therapy
6. Life expectancy <1 year
7. Participation in another trial related to β-blockers or other anti-anginal drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8500 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of time to first all-cause death, non-fatal MI, or hospitalization for resuscitated cardiac arrest, unstable angina requiring urgent revascularization or heart failure over an estimated four years | 4 years post randomization
  Composite of time to first all-cause death, non-fatal MI, or hospitalization for resuscitated cardiac arrest, unstable angina requiring urgent revascularization or heart failure over an estimated four years

SECONDARY OUTCOMES:
individual components of the primary objective (including all-cause death, non-fatal MI, or hospitalization for resuscitated cardiac arrest, unstable angina requiring urgent revascularization or HF) | 4 years post randomization
  individual components of the primary objective (including all-cause death, non-fatal MI, or hospitalization for resuscitated cardiac arrest, unstable angina requiring urgent revascularization or HF)
stroke | 4 years post randomization
  stroke
angina related quality of life | 4 years post randomization
  angina related quality of life as measured by the Seattle Angina Questionnaire
sexual function | 4 years post randomization
  sexual function as measured by the IIEF-5 and FSFI
new onset diabetes | 4 years post randomization
  new onset diabetes
drug withdrawal | 4 years post randomization
  stop/re-start dates
health care costs in each arm | 4 years post randomization
  health care costs in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No